CLINICAL TRIAL: NCT03332030
Title: Development of Stem Cell Lines in Children With Neurofibromatosis Type 1 and Tumors of the Central Nervous System
Brief Title: Stem Cells in NF1 Patients With Tumors of the Central Nervous System
Status: Withdrawn | Type: Observational
Why Stopped: Suspended due to cessation of funding
Sponsor: Roger Packer (Other)
Responsible Party: Sponsor-Investigator, Roger Packer, Senior Vice President, Center for Neuroscience & Behavioral Health, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: Pro00006360
Record Dates: First submitted 2017-06-26; First posted 2017-11-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Neurofibromatosis Type 1; Tumors of the Central Nervous System
MeSH Terms: conditions — Neurofibromatosis 1; Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 20 ml of whole blood obtained to develop stem cell lines
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Collection of Stem Cells — One time collection of a 20 ml blood sample

SUMMARY:
Objectives 1. Establish an induced pluripotent stem cell (iPSC) bank for phenotypically well-characterized patients with NF1.

2. Develop isogenic NF1 wild-type (NF1+/+), NF1 heterozygous (NF1+/-) and NF1 homozygous (NF1-/-) iPSC lines from individual patients using CRISPR/CAS9 technology.

3. Differentiate and characterize disease-relevant brain cells such as excitatory and inhibitory neurons, astrocytes and oligodendrocytes from patient-specific iPSC lines.

4. Screen and identify the drug(s) that can reverse or alleviate the disease phenotypes.

DETAILED DESCRIPTION:
Hypothesis: Subjects with NF1 and central nervous system tumors who have aggressive lesions (including, but not limited to optic pathway gliomas) and/or those with tumors causing neurologic (including visual) morbidity will manifest unique differences in their stem cells and stem cell-derived differentiated cells compared to patients with NF1 and central nervous system tumors who have less aggressive disease and/or those with tumors causing minimal to no morbidity.

Background and Significance: Optic pathway gliomas (OPGs) are low-grade astrocytic tumors primarily involving the optic nerve, chiasm and tracts that occur mainly in children. Nearly 20% of children with Neurofibromatosis type 1 (NF1) will develop OPGs, although less than half will develop vision loss from their tumor.1 These tumors have excellent survival outcomes, making vision loss the primary morbidity in these patients. Furthermore, OPGs are inherent to the visual pathway, therefore they are rarely, if ever biopsied. This paucity of OPG tissue limits our ability to clarify the biologic differences between OPGs that cause vision loss and those that do not. Low-grade astrocytic gliomas in the other regions of the brain including the hypothalamus, brainstem and cerebellum can also be found in a subset of children associated with NF1. These NF1-associated brain tumors can progress and also grow at variable rates and may cause neurologic dysfunction ranging from severe compromise to little or no symptomality.

This study seeks to develop stem cells lines in children with NF1-related tumors in the central nervous system (the optic nerve and those from other brain sites). Stem cells from these subjects will provide a critical insight into the mechanisms responsible for tumor progression and symptoms associated with the central nervous system, accelerating the identification of therapeutic targets.

Preliminary Studies: Three recent research developments make it possible to develop a patient-specific disease model in a dish (so-called "human disease model in dish") and to study induced pluripotent stem cell (iPSC)-derived disease relevant cells in an isogenic background. First, embryonic stem cell (ESC)-like cells, also known as induced pluripotent stem cell or iPSC, can be generated from skin or blood cells in adult patients. Second, recent research efforts have started to develop culture protocols that differentiate iPSCs into a variety of cell types in the central and peripheral nervous system (CNS and PNS), which are affected in NF1 patients. Third, the CRISPR/CAS9 technology allows to genetically edit the specific disease genes either by repairing the existing mutant genes or creating new mutations. In order to position at the forefront of NF1 research, it will be important for the Gilbert Family Neurofibromatosis Institute (GFNI) at the Children's National Medical Center to explore these recent exciting research developments, to systematically develop patient-specific human NF1 disease models, and to provide a tool for drug screening and evaluation on the individual NF patients.

Design and Methods:

3.1 Study Design Cross-sectional collection of NF1 subjects with tumors in the central nervous system as documented by MRI.

3.2 Study Visits Subjects will have only one visit to collect the blood sample.

3.3 Study Procedures 3.31 Blood Draw Subjects have 20 ml of whole blood drawn during either 1)their sedation for their clinically indicated MRI (IV already being placed for clinical purpose) or through the outpatient laboratory.

3.32 Stem Cell Processing Blood collected will be immediately transferred to the stem cell facility at the National Institutes of Health for processing of the specimens in order to develop stem cell lines.

3.33 Demographics We will collect the subject's age, gender, race, ethnicity, location of tumors in the central nervous system on MRI, history of vision loss and other neurological deficits.

3.34 Statistical Analysis As a first step to establish a stem cell library from a specific population of NF1 children with nervous system tumors, we will not need statistical analysis at this stage.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of any age
* Confirmed diagnosis of NF1
* Willingness to submit blood sample and collect clinical history
* MRI documentation confirming tumor location in the central nervous system.
* For study group d, "Non-NF1 full sibling for control purposes" subject must be a full sibling of a patient with confirmed diagnosis of NF1 and willing to submit blood sample and collect clinical history.

Exclusion Criteria:

* Does not have diagnosis of NF1 and CNS Tumor
* Does not have full-sibling with NF1 and CNS Tumor diagnosis (for unaffected sibling cohort)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. NF1 with tumors in the central nervous system, asymptomatic (normal vision), not treated
  2. NF1 with tumors in the central nervous system, symptomatic, not treated/impending treatment
  3. NF1 with tumors in the central nervous system, symptomatic, treatment completed > 2 years ago.
  4. Non-NF1 full sibling for control purposes
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The identity of mutations in NF1 genes will be measured. | June 2019
  The stem-cell characteristics of patient-derived induced pluripotent stem cell (iPSC) lines will be measured and reported.

SECONDARY OUTCOMES:
The iPS cell lines with NF1 mutations will be engineered to inactivate the remaining NF1 wild-type or fix the mutant allele using CRISPR/CAS9 technology. | June 2019
  The status of NF1 gene will be measured for the isogenic NF1 wild-type (NF1+/+), NF1 heterozygous (NF1+/-) and NF1 homozygous (NF1-/-) iPSC lines. The stem cell characteristics of isogenic NF1 iPSC lines will be measured.
Measure neuronal characteristics of neurons derived from iPSC lines. | June 2019
  Differentiate between and characterize the disease-relevant brain cells (excitatory and inhibitory interneurons, astrocytes, and oligodendrocytes) of the patient's iPSC (induced pluripotent stem cell) lines.
Measure glial properties of glia derived from iPSC lines. | June 2019
  After characterizing the disease-relevant brain cells (excitatory and inhibitory neurons, astrocytes, and oligodendrocytes) from patient-specific iPSC lines, screen and identify the drug(s) that can reverse or alleviate the specific disease phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Packer, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States